CLINICAL TRIAL: NCT00231608
Title: The Safety and Efficacy of Topiramate in Male Patients With Abdominal Obesity: A 6-Month Double-Blind, Randomized, Placebo-Controlled Study With a 6-Month Open-Label Extension
Brief Title: A Study of Safety and Efficacy of Topiramate in Male Patients With Abdominal Obesity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR003724
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-04

CONDITIONS: Obesity
Keywords: Obesity; Abdominal Obesity; Visceral Fat; Subcutaneous Fat; Dislipidemia; Hypertension; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Obesity; Obesity, Abdominal; Hypertension; Diabetes Mellitus, Type 2 | interventions — Topiramate

INTERVENTIONS:
Drug: topiramate

SUMMARY:
The purposes of this study are to compare the effects of Topiramate and placebo on abdominal visceral fat accumulation at 6 months and to evaluate the safety of Topiramate for up to 12 months of continued treatment in male patients with abdominal obesity.

DETAILED DESCRIPTION:
Topiramate is not approved for the treatment of obesity. This study is a 6-month randomized, double-blind placebo-controlled study, followed by a 6-month open-label extension study to evaluate the effect of Topiramate on abdominal visceral fat accumulation, a clinical surrogate known to be associated with the complications of obesity such as increased incidence of Type 2 diabetes mellitus, hypertension, and dyslipidemia, and their associated morbidities. Patients will be randomized to receive either daily Topiramate or placebo. Effectiveness will be measured by multiple parameters such as abdominal visceral fat (assessed by computed tomography), total and subcutaneous abdominal fat, body composition, body weight, body mass index, glucose tolerance, lipid profile, blood pressure, Topiramate plasma concentration, or 24 hours energy expenditure (selected patients). Safety evaluation (adverse events, vital signs, 12-lead ECG, clinical laboratory tests) will be conducted throughout the study. The study hypothesis is that Topiramate is effective in reducing abdominal visceral fat in male patients and well tolerated. After the initial 12-week titration phase, patients will receive either Topiramate (200mg twice daily or the maximum dose tolerated) or placebo by mouth for 6-months. Then, patients will receive Topiramate (200mg twice daily or the maximum tolerated dose) for 6-months during the open-label phase.

ELIGIBILITY:
Inclusion Criteria:

* BMI >= 27 and =< 40
* a waist circumference >= 100 cm (39.4 inches)
* Baseline weight must be stable (varying no more than 4 kg (8.8 lbs)) for at least two months prior to enrollment
* Must be sedentary (less than one session of continuous moderate physical activity of 30 min/week)
* Must have blood lipid disorder
* Must be non-smokers

Exclusion Criteria:

* Patients with endocrine disease or other physical causes of obesity
* Patients with significantly abnormal hepatic liver function tests or renal disease
* History of schizophrenia, psychotic, or major affective disorder
* History of epilepsy
* History of eating disorders
* History of any other significant medical conditions

Ages: 25 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 1998-12; Study Completion 2002-01 (Actual)

PRIMARY OUTCOMES:
The mean change from baseline to Month 6 in abdominal visceral fat as assessed by computed tomography; the safety of Topiramate for up to 12 months of continued treatment in male subjects with abdominal obesity.

SECONDARY OUTCOMES:
Mean change and percent change in body weight, and mean change in total abdominal fat, subcutaneous abdominal fat, body composition, and body mass index from baseline to Month 6.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A Study of Safety and Efficacy of Topiramate in Male Patients with Abdominal Obesity — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=540&filename=CR003724_CSR.pdf